CLINICAL TRIAL: NCT00515424
Title: A Multicenter, Randomized, Placebo-Controlled, Latanoprost-Controlled, Parallel Group Study to Assess the Tolerability, Safety and Efficacy of RKI983 Ophthalmic Solution Given Twice a Day Over One Week in Patients With Primary Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Tolerability, Safety and Efficacy of RKI983 Eye Drops in Subjects With Primary Open Angle Glaucoma and Ocular Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRKI983A2101
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Ocular Hypertension; RKI983; Primary Open Angle Glaucoma and Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Glaucoma, Open-Angle

INTERVENTIONS:
Drug: RKI983

SUMMARY:
This study will evaluate the tolerability and safety of RKI983 ophthalmic solution and explore the effect of the compound on intraocular pressure in subjects with ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ≥18 years of age, with primary open angle glaucoma and ocular hypertension
* Females must be post-menopausal or surgically sterile

Exclusion Criteria:

* Other types of glaucoma
* Eye pressure lowering surgeries
* A history of or current eye conditions or medical problems that would prohibit the use of an investigational drug

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2007-07

PRIMARY OUTCOMES:
Rates of adverse events and serious adverse events, as well as changes in ophthalmic evaluations, laboratory values, ECGs and vital signs over period of 7 days treatment.

SECONDARY OUTCOMES:
Change in ocular hypertension from Baseline to Day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Independent Central IRB
Locations (5):
- United States (5):
  - Artesia, California
  - Rochester, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Houston, Texas